CLINICAL TRIAL: NCT06854159
Title: A Phase 2 Study of Odronextamab in Relapsed/ Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL) Before and After Chimeric Antigen Receptor (CAR) T-Cell Therapy
Brief Title: Odronextamab for the Treatment of Relapsed and Refractory Diffuse Large B-cell Lymphoma Before and After Chimeric Antigen Receptor T-cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC310; NCI-2025-00900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC310 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); UCHMC2329 (Other: UC Hematologic Malignancies Consortium); R1979-HM-2494 (Other Grant/Funding Number: Regeneron)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (odronextamab, CAR T-cell therapy) (Experimental): Patients receive odronextamab IV over 1-4 hours on days 1, 2, 8, 9, 15, and 16 of cycle 1, on days 1, 8, and 15 of cycles 2-4 then on days 1 and 15 of subsequent cycles until achievement of durable CR. Cycles repeat every 21 days in the absence of durable CR, disease progression, or unacceptable toxicity. Patients with durable CR for ≥ 9 months may then receive odronextamab IV over 1-4 hours on day 1 of each subsequent cycle. These cycles repeat every 28 days for up to a total of 2 years in the absence of disease progression or unacceptable toxicity. Patients receive SOC CAR T-cell therapy if disease assessment shows less than a CR after cycle 4, or after cycle 5 if disease assessment shows PD any time after cycle 5.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Biological: Odronextamab

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Receive CAR T-cell therapy
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Biological: Odronextamab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody REGN1979; REGN1979; WHO 11035

SUMMARY:
This phase II trial tests how well odronextamab works before and after standard of care (SOC) chimeric antigen receptor (CAR) T-cell therapy in treating patients with diffuse large B-cell lymphoma (DLBCL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). CAR-T cell therapy is the SOC treatment most patients receive when other treatments have failed. CAR-T cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Odronextamab is a monoclonal antibody that is called bispecific, as it individually targets 2 cell proteins, CD20 and CD3. Proteins are part of each cell in the body, which work together like little machines for the cell to function. CD20 is a protein that is found on the surface of both normal B-cells and B-cells that make up certain cancers, like DLBCL. CD3 is a protein that is found on the surface of T cells. T-cells and normal B-cells are types of white blood cells in the body and are a part of the immune system that fights infections. Odronextamab is designed to help T-cells find and kill the B-cells including the cancer cells in DLBCL. Giving odronextamab before and after CAR T-cell therapy may improve response in patients with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess anti-tumor activity of odronextamab + CAR T-cell therapy in in patients with relapsed or refractory (R/R) DLBCL.

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of odronextamab + CAR T-cell therapy in patients with R/R DLBCL.

II. To further assess anti-tumor activity of odronextamab + CAR T-cell therapy in patients with R/R DLBCL.

OUTLINE:

Patients receive odronextamab intravenously (IV) over 1-4 hours on days 1, 2, 8, 9, 15, and 16 of cycle 1, on days 1, 8, and 15 of cycles 2-4 then on days 1 and 15 of subsequent cycles until achievement of durable complete response (CR). Cycles repeat every 21 days in the absence of durable CR, disease progression, or unacceptable toxicity. Patients with durable CR for ≥ 9 months may then receive odronextamab IV over 1-4 hours on day 1 of each subsequent cycle. These cycles repeat every 28 days for up to a total of 2 years in the absence of disease progression or unacceptable toxicity. Patients receive SOC CAR T-cell therapy if disease assessment shows less than a CR after cycle 4, or after cycle 5 if disease assessment shows progressive disease (PD) any time after cycle 5. Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and blood sample collection, positron emission tomography (PET)/computed tomography (CT) or CT throughout the study. Patients may also undergo CT of the brain at screening.

After completion of study treatment, patients are followed up at 30 days then every 4 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 at the time of consent
* Patients must have histologically or cytologically confirmed relapsed/ refractory (R/R) diffuse large B-cell lymphoma (DLBCL); transformed follicular lymphoma patients are eligible
* Patients must have failed at least 2 prior therapies
* Life expectancy ≥ 3 months
* Candidate for any Food and Drug Administration (FDA)-approved chimeric antigen receptor (CAR) T cell therapy as per institutional guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 50%)
* Leukocytes ≥ 2,500/µL
* Absolute neutrophil count ≥ 1,000/µL or > 500/µL for patients with bone marrow involvement

  * A participant may not have received granulocyte colony stimulating factor within 2 days prior to first dose of odronextamab in order to meet the absolute neutrophil count (ANC) eligibility criterion
* Platelets ≥ 50,000/µL or ≥ 25,000/µL for patients with bone marrow involvement

  * A patient may not have received platelet transfusion therapy within 2 days prior to first dose of odronextamab in order to meet the platelet eligibility criterion
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)

  * NOTE: patients with known Gilbert disease who have serum bilirubin level ≤ 3 x institutional ULN may be enrolled. Patients with known Gilbert syndrome will be excluded if the total bilirubin value is > 4 x ULN
  * Irrespective of the presence of lymphoma infiltration of the liver, a participant with an aspartate aminotransferase (AST) > 3 x ULN and/or alanine aminotransferase (ALT) > 3 x ULN concurrent with a total bilirubin > 1.5 x ULN will be excluded
* AST(serum glutamic oxaloacetic transaminase [SGOT])/ALT(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN (AST and/or ALT ≤ 5 x ULN for patients with liver involvement)

  * Irrespective of the presence of lymphoma infiltration of the liver, a participant with an AST > 3 x ULN and/or ALT > 3 x ULN concurrent with a total bilirubin > 1.5 x ULN will be excluded
* Creatinine clearance ≥ 30 mL/min/1.73 m^2 by Cockcroft-Gault
* Hemoglobin ≥ 8 g/dL or ≥ 7 g/dL for patients with bone marrow involvement

  * NOTE: Growth factor or transfusion support is allowed as per treating physician's discretion
* Alkaline phosphatase 2.5 x ULN (≤ 5 x ULN for patients with documented liver involvement or bone metastases)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN

  * NOTE: This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose
* Cardiac ejection fraction > 50% by echocardiogram or multigated acquisition (MUGA) scan
* Serum creatinine ≤ 1.5 x ULN, or calculated creatinine clearance by Cockcroft Gault formula ≥ 50 mL/min
* For participants infected with HIV:

  * No history of AIDS-defining conditions other than lymphoma or history of CD4+ T-cells below 200/mm^3 prior to beginning combination antiretroviral therapy (ART)
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
  * At time of study entry CD4+ T-cells must have recovered from prior lymphoma therapy to ≥ 250/mm^3
  * At the time of study entry, the HIV viral load must be undetectable by standard laboratory assay
  * During prior lymphoma therapy, patients must not have experienced documented infections attributed to the HIV+ status
  * No history of non-adherence to ART and willing to adhere to ART while on study
  * Antiretroviral drugs with overlapping or similar toxicity profiles as study agents not allowed
* People with hepatitis B or C on suppressive therapy with a negative viral load and no evidence of hepatic damage are eligible
* People of child-bearing potential and reproductive partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months (180 days) after the last dose of study agent. Egg and sperm donation is prohibited during the study and for 6 months after the last dose of study agent
* Willing and able to provide informed consent

Exclusion Criteria:

* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she/they were to participate in the study or confounds the ability to interpret data from the study as determined by the study principal investigator (PI) or enrolling physician
* Known involvement by primary central nervous system (CNS) lymphoma or known uncontrolled involvement by non-primary CNS non-Hodgkin lymphoma (NHL) at the time of study entry
* Known history (within last 12 months) of or current relevant CNS pathology, such as:

  * Epilepsy, seizure, paresis, aphasia, apoplexy, severe brain injury, cerebellar disease, organic brain syndrome, psychosis, cerebrovascular stroke or
  * Evidence for presence of inflammatory lesions and/or vasculitis on cerebral magnetic resonance imaging (MRI)
* Another active malignancy (aside from B-cell NHL) in the past 5 years, with the following exceptions: non-melanoma skin cancer that has undergone potentially curative therapy, in situ cervical carcinoma, or any other tumor that has been deemed to be effectively treated with definitive local control and with curative intent as per treating investigator
* Evidence of any active infection (bacterial, viral, fungal, mycobacterial, parasitic, or other) at study enrollment or within 2 weeks of study enrollment, if requiring ongoing treatment and/or has the potential to cause disseminated disease or severe infection upon immunosuppression. There should be evidence that the infection has cleared or is well controlled by start of study therapy
* Active COVID-19 infection
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)

  * Participants with HIV who have controlled infection (undetectable viral load and CD4 count above 350 cells/µL either spontaneously or on a stable antiviral regimen) are permitted.
  * Participants who are hepatitis B surface antigen positive or who are hepatitis B core antibody positive should undergo evaluation by a specialist and be considered to have controlled infection (serum hepatitis B virus deoxyribonucleic acid [DNA] polymerase chain reaction [PCR] that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) before they are permitted onto study
  * Participants who are HCV antibody positive who have controlled infection (undetectable HCV ribonucleic acid [RNA] by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted
* Cytomegalovirus (CMV) infection as noted by detectable levels on peripheral blood polymerase chain reaction (PCR) assay. Patients who show detectable levels of CMV at screening will need to be treated with appropriate antiviral therapy and demonstrate at least 2 undetectable levels of CMV by PCR assay (at least 7 days apart) before being re-considered for eligibility
* Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone/prednisolone or anti-inflammatory equivalent within 72 hours of start of assigned treatment
* Recent major surgery (within 4 weeks prior to the start of study treatment)
* Standard radiotherapy within 14 days of first administration of study treatment
* Prior organ transplantation
* Administration of live vaccination within 28 days of study first dose
* Use of any other experimental drug or therapy within 28 days (or 5 half-lives of the drug, whichever is shorter) of initiating study treatment
* Concurrent use of other anti-cancer treatments except for certain therapeutics (e.g., maintenance hormonal-based therapy) per the treating physician's discretion
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* Pregnancy or lactation
* Known allergic reactions or hypersensitivity to allopurinol, rasburicase, or compounds of similar chemical or biological components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | From first dose through completion of 5 cycles (cycle length = 21 days for cycles 1-4 and 14 days for cycle 5) of odronextamab and chimeric antigen receptor (CAR) T cell infusion
  Will be assessed by Lugano 2014. Will calculate the uniformly minimum variance unbiased estimator, p-value, and confidence intervals for CRR. The calculation will be performed using R clinfun package.

SECONDARY OUTCOMES:
Number of participants experiencing treatment-related adverse events (AEs) | From first dose through 30 days post last odronextamab dose
  Will be classified by severity, and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The proportion of subjects experiencing AEs, serious AEs, and treatment delays will be summarized. All AEs will be listed, documenting the course, outcome, severity, and relationship to the study treatment. Incidence rates of AEs and the proportion of subjects prematurely withdrawn from the study due to AEs will be reported.
Number of participants with progression-free survival | From the date of first odronextamab dose until the first occurrence of disease progression, or death from any cause, whichever occurs earlier, assessed up to 2 years
  Will be summarized using Kaplan-Meier methodology using 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals (CIs), as well as number and percentage of censored observations.
Objective response rate | From first dose to up to 2 years post last odronextamab dose
  Will be assessed by Lugano 2014. Data will be presented using descriptive statistics. Tabulations will be produced for appropriate disposition, demographic, baseline, efficacy, and safety parameters. For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) of the parameter will be presented, as well as 2-sided 95% CIs, unless stated otherwise. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.
Number of minimal residual disease (MRD) negative targets detected | After cycle 4 (pre-CAR T-cell therapy) and 2 cycles post CAR T cell infusion (cycle length = 21 days for cycles 1-4 and 14 days for subsequent cycles)
  Will use circulating tumor-derived deoxyribonucleic acid testing. Data will be presented using descriptive statistics. Tabulations will be produced for appropriate disposition, demographic, baseline, efficacy, and safety parameters. For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) of the parameter will be presented, as well as 2-sided 95% CIs, unless stated otherwise. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States